CLINICAL TRIAL: NCT06557135
Title: Brachial vErsus Femoral Access for carotId Artery sTenting: a Multicenter Randomized Clinical Trial (BEFIT)
Brief Title: Brachial Versus Femoral Access for Carotid Artery Stenting
Acronym: BEFIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Liu Sheng, Chief Physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-SR-534
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Carotid Artery Stenosis Without Infarction (Disorder); Ischemic Stroke
Keywords: Brachial Artery; Femoral Artery; Carotid Artery Stenting; Carotid Stenosis
MeSH Terms: conditions — Ischemic Stroke; Carotid Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the brachial group (Experimental): Patients with carotid artery stenosis will be randomly selected for carotid artery stenting via the brachial artery access.
  Interventions: Procedure: Carotid Artery Stenting (CAS)
- the femoral group (Active Comparator): Patients with carotid artery stenosis will be randomly selected for carotid artery stenting via the femoral artery access.
  Interventions: Procedure: Carotid Artery Stenting (CAS)

INTERVENTIONS:
Procedure: Carotid Artery Stenting (CAS) — CAS involves inserting a catheter or tube into an artery in the brachial or the femoral, and then threading the catheter through the arteries of the body to the location of the stenosis within the carotid artery in the neck. A stent is then placed in the stenosis and holds the artery open.

SUMMARY:
Study purpose:

A multicenter, prospective and randomized study is planned to compare the clinical outcomes of carotid artery stenting via brachial artery access and femoral artery access.

Eligible participants will be randomly assigned 1:1 to the brachial artery group or the femoral artery group.

Primary endpoint: surgical success rate.

Secondary endpoints:

1. Operation time (time from first arterial puncture to last angiography)
2. Serious adverse events (SAE) within 90 days;
3. Access puncture complications;

DETAILED DESCRIPTION:
With the improvement of treatment concepts and the continuous innovation of interventional devices/interventional technologies, neurointervention has become the preferred treatment method for many cerebrovascular diseases. Among them, the femoral artery is the most commonly used access, because the femoral artery is superficial, easy to touch, and the relatively large vessel diameter allows most neurointerventional surgeries to proceed smoothly. However, the femoral artery access also has the disadvantages of long bed rest time, exposure to private parts, and prolonged hospitalization.

Thanks to the great success of radial artery access in cardiac intervention, radial artery access is increasingly being used in neurointervention. However, due to the thin radial artery, there is a significantly increased risk of complications (radial artery spasm, radial artery occlusion) during large-cavity nerve intervention, and the operation time is significantly prolonged. Therefore, the overall proportion of neurointerventional treatment via radial artery access in clinical practice is less than 12%.

As the superior vascular trunk of the radial artery, the brachial artery has a larger diameter and is theoretically more suitable to replace the radial artery for large-bore intervention. Anatomically, the brachial artery is superficial and easy to touch in the antecubital fossa, and there are no important vessels and nerves in front of the blood vessel, and the posterior is the distal humeral platform, which is easy for brachial artery puncture and postoperative compression hemostasis. Studies have shown that thrombectomy for cerebral artery occlusion and carotid artery stent placement can be safely performed through the brachial artery. However, current studies are based on single-center small sample studies, and there is still a lack of large-sample randomized controlled trials to verify the safety and effectiveness of neurointervention via the brachial artery.

This study intends to conduct a multicenter, prospective, and randomized study to compare the clinical results of carotid artery stent placement via the brachial and femoral artery access.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stenosis at the origin of the carotid artery with indications for neuro-interventional treatment (symptomatic stenosis >50%; asymptomatic stenosis >70%)
* Aged 18 or above
* With palpable brachial and femoral arteries
* The patient or his/her agent understands the purpose and needs of this study and signs the informed consent

Exclusion Criteria:

* Symptomatic stenosis or occlusion of multiple vessels at the same time
* Intravascular intervention for multiple vessel lesions at the same time
* Ischemic stroke within the past 2 weeks
* Any active bleeding, severe anaemia, or coagulation disorder. At least one of the following laboratory tests must be met: haemoglobin < 10g/dL, or platelet count < 100,000 /μ L, or unadjusted INR >1.5, or PT exceeds the upper limit of normal by 1 minute or heparin-induced thrombocytopenia
* A large-area cerebral infarction stroke on the same side with sequelae may affect the judgment of the study endpoint
* A history of cerebral hemorrhage in the past six months
* Any condition that may interfere with digital subtraction angiography (DSA) or cause unsafe percutaneous arterial access Participating in other clinical trials, in the research stage or follow-up stage
* Contraindications to cerebral angiography, such as allergy to iodine contrast agents and renal insufficiency
* Unable to understand or sign the informed consent form
* Severe functional damage to important organs, assessed by clinical physicians to have high surgical risks and intolerant of interventional surgery
* Baseline modified Rankin scale greater than or equal to 2
* Expected survival is less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful rate of CAS | 24 hours
  Successful carotid artery stenting (CAS) is defined as access devices can be established, interventional devices can reach the lesion site, operations such as distal brain protection device release, balloon expansion and stent implantation, withdrawal protection device can be completed successfully, and residual stenosis < 30%.

SECONDARY OUTCOMES:
Procedure time | 24 hours
  time from first arterial puncture to last angiography
Serious adverse events (SAE) | 90 days
  SAEs related to operation and device are defined as those related to operation procedure and device determined by investigators. Includes the incidence of death, new-onset stroke, or severe haemorrhage events within 90 days post-procedure, et al.
Access puncture complications | 90 days
  Hematoma at access puncture site, pseudoaneurysm, arteriovenous fistula, symptomatic severe stenosis/occlusion

OTHER OUTCOMES:
X-ray exposure | 24 hours
  X-ray exposure is defined as the duration and equivalent of X-ray exposure recorded by the DSA machine during operation.
Access conversion | 24 hours
  If the randomized access was not successfully completed, switched to other access
Degree of patient-reported comfort | 24 hours
  The comfort scale adopts the simplified General Comfort Questionnaire (GCQ）developed by nursing expert Kolcaba. The scale is scored by level 1 to 4 Likert scale, with a score range of 28-112 points. The lowest score is 28 points and the highest score is 112 points. The higher the score, the higher the comfort. A total score of < 60 is low comfort, a total score of 60-90 is moderate comfort, and a total score of > 90 is high comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Liu, Professor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sousa-Uva M, Neumann FJ, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur J Cardiothorac Surg. 2019 Jan 1;55(1):4-90. doi: 10.1093/ejcts/ezy289. No abstract available. PMID 30165632
- [Background] Kenawy AE, Tekle W, Hassan AE. Improved Fluoroscopy and Time Efficiency with Radial Access for Diagnostic Cerebral Angiography. J Neuroimaging. 2021 Jan;31(1):67-70. doi: 10.1111/jon.12807. Epub 2020 Nov 16. PMID 33191571
- [Background] Stone JG, Zussman BM, Tonetti DA, Brown M, Desai SM, Gross BA, Jadhav A, Jovin TG, Jankowitz B. Transradial versus transfemoral approaches for diagnostic cerebral angiography: a prospective, single-center, non-inferiority comparative effectiveness study. J Neurointerv Surg. 2020 Oct;12(10):993-998. doi: 10.1136/neurintsurg-2019-015642. Epub 2020 Jan 22. PMID 31974282
- [Background] Haussen DC, Nogueira RG, DeSousa KG, Pafford RN, Janjua N, Ramdas KN, Peterson EC, Elhammady MS, Yavagal DR. Transradial access in acute ischemic stroke intervention. J Neurointerv Surg. 2016 Mar;8(3):247-50. doi: 10.1136/neurintsurg-2014-011519. Epub 2015 Jan 5. PMID 25561585
- [Background] Montorsi P, Galli S, Ravagnani MP, Teruzzi G, Calligaris G, Gili S, Caputi L, Troiano S, Del Maso R, Trabattoni D. Transradial/brachial carotid artery stenting with proximal protection: technical instructions, acute results and long-term outcomes. Minerva Cardiol Angiol. 2022 Dec;70(6):765-777. doi: 10.23736/S2724-5683.22.06223-8. Epub 2022 Dec 15. PMID 36519647
- [Background] Lu CJ, Lin YH, Chu HJ, Tang SC, Lee CW. Safety and efficacy of the transbrachial approach for endovascular thrombectomy in patients with acute large vessel occlusion stroke. J Formos Med Assoc. 2021 Jan;120(1 Pt 3):705-712. doi: 10.1016/j.jfma.2020.08.002. Epub 2020 Aug 17. PMID 32819794
- [Background] Starke RM, Snelling B, Al-Mufti F, Gandhi CD, Lee SK, Dabus G, Fraser JF; Society of NeuroInterventional Surgery. Transarterial and transvenous access for neurointerventional surgery: report of the SNIS Standards and Guidelines Committee. J Neurointerv Surg. 2020 Aug;12(8):733-741. doi: 10.1136/neurintsurg-2019-015573. Epub 2019 Dec 9. PMID 31818970
- [Background] Naylor R, Rantner B, Ancetti S, de Borst GJ, De Carlo M, Halliday A, Kakkos SK, Markus HS, McCabe DJH, Sillesen H, van den Berg JC, Vega de Ceniga M, Venermo MA, Vermassen FEG, Esvs Guidelines Committee, Antoniou GA, Bastos Goncalves F, Bjorck M, Chakfe N, Coscas R, Dias NV, Dick F, Hinchliffe RJ, Kolh P, Koncar IB, Lindholt JS, Mees BME, Resch TA, Trimarchi S, Tulamo R, Twine CP, Wanhainen A, Document Reviewers, Bellmunt-Montoya S, Bulbulia R, Darling RC 3rd, Eckstein HH, Giannoukas A, Koelemay MJW, Lindstrom D, Schermerhorn M, Stone DH. Editor's Choice - European Society for Vascular Surgery (ESVS) 2023 Clinical Practice Guidelines on the Management of Atherosclerotic Carotid and Vertebral Artery Disease. Eur J Vasc Endovasc Surg. 2023 Jan;65(1):7-111. doi: 10.1016/j.ejvs.2022.04.011. Epub 2022 May 20. No abstract available. PMID 35598721
- [Background] Kendrick DB, Strout TD. The minimum clinically significant difference in patient-assigned numeric scores for pain. Am J Emerg Med. 2005 Nov;23(7):828-32. doi: 10.1016/j.ajem.2005.07.009. PMID 16291435
- [Background] Heck D, Jost A, Howard G. Stenting the carotid artery from radial access using a Simmons guide catheter. J Neurointerv Surg. 2022 Feb;14(2):169-173. doi: 10.1136/neurintsurg-2020-017143. Epub 2021 Feb 25. PMID 33632887
- [Background] Jaroenngarmsamer T, Bhatia KD, Kortman H, Orru E, Krings T. Procedural success with radial access for carotid artery stenting: systematic review and meta-analysis. J Neurointerv Surg. 2020 Jan;12(1):87-93. doi: 10.1136/neurintsurg-2019-014994. Epub 2019 Jun 14. PMID 31201288
- [Background] Dossani RH, Waqas M, Monteiro A, Cappuzzo JM, Almayman F, Snyder KV, Levy EI, Siddiqui AH, Davies JM. Use of a sheathless 8-French balloon guide catheter (Walrus) through the radial artery for mechanical thrombectomy: technique and case series. J Neurointerv Surg. 2022 May;14(5):neurintsurg-2021-017868. doi: 10.1136/neurintsurg-2021-017868. Epub 2021 Aug 24. PMID 34429347
- [Background] Hernandez D, Requena M, Olive-Gadea M, de Dios M, Gramegna LL, Muchada M, Garcia-Tornel A, Diana F, Rizzo F, Rivera E, Rubiera M, Pinana C, Rodrigo-Gisbert M, Rodriguez-Luna D, Pagola J, Carmona T, Juega J, Rodriguez-Villatoro N, Molina C, Ribo M, Tomasello A. Radial Versus Femoral Access for Mechanical Thrombectomy in Patients With Stroke: A Noninferiority Randomized Clinical Trial. Stroke. 2024 Apr;55(4):840-848. doi: 10.1161/STROKEAHA.124.046360. Epub 2024 Feb 1. PMID 38299334